CLINICAL TRIAL: NCT05126914
Title: Multicentre Real-life Follow-up Study of Rare Epileptic Syndromes in Children and Adolescents
Acronym: EPIRARE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Orphelia Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: P210776
Record Dates: First submitted 2021-10-22; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Epilepsy; West Syndrome; Dravet Syndrome
MeSH Terms: conditions — Epilepsy; Spasms, Infantile; Epilepsies, Myoclonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rare epilepsies as a whole account for 20-30% of epilepsies, but knowledge about prognostic factors is currently limited. This means that it is difficult to provide adequate information to families at diagnosis and during follow-up. Prognostic factors are also important for management as they can have an impact on the patient's outcome (time to intervention, choice of one molecule over another, etc.). Finally, few treatments are currently available for these epilepsies. One of the limitations to the development of treatments is the lack of real life data as it is difficult to create reliable primary endpoints such as the rate of patients becoming seizure free naturally compared to a therapeutic intervention.

The aim of this real-life study is to evaluate the response to treatment as well as to see the evolution of cognitive and psychiatric comorbidities. As explained above, there are very few randomised trials except for 3 rare epilepsies (infantile spasm syndrome, Dravet syndrome, Lennox-Gastaut syndrome). This has led to the virtual absence of management recommendations, including for the three syndromes mentioned above, where attempts at treatment algorithms have been proposed, although these have not been able to be considered as evidence-based recommendations.

As a result, there is some diversity in the management of rare epilepsies from one centre to another. However, this diversity in management can be an asset in a real-life study. This will make it possible to compare different management methods, both in terms of seizure control and medium-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis for rare epilepsy (based on ORPHA codes)
* holders of parental authority not opposed
* Be followed in one of the declared centers of the study

Exclusion Criteria:

* opposition from the holders of parental authority or the patient

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population studied in this work will be a pediatric population: from birth to the end of adolescence. There is no limitation in the epileptic syndromes provided that it is a rare epilepsy according to the waxers with a prevalence of 1 in 2000. As mentioned here on several occasions, there is little data on it. efficacy of treatments and the outcome of rare epilepsies. A fairly wide opening on the syndromes to be included will make it possible to collect data without being limited to those which are the subject of the most frequent publications and therefore provide data not available to date.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
rate of decrease in epileptic seizures | 5 years
  rate of decrease in epileptic seizures according to the treatments used based on the seizure calendar kept by the parents as part of the current care.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane AUVIN, Pr, Study Director — Hopital Robert Debré - Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Robert Debré - Neurologie, Paris, France

IPD SHARING:
Plan to Share IPD: No
non available